CLINICAL TRIAL: NCT05514106
Title: Myocardial 123I-MIBG Scintigraphy in Aging and Neurodegenerative Disease
Brief Title: MIBG in Aging and Neurologic Disorders
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bradley Boeve, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-012740
Record Dates: First submitted 2022-08-23; First posted 2022-08-24 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Lewy Body Disease; Dementia; Parkinsonism; Mild Cognitive Impairment; REM Sleep Behavior Disorder
Keywords: REM Sleep without atonia; Normal Neurologic functioning
MeSH Terms: conditions — Lewy Body Disease; Dementia; Parkinsonian Disorders; Cognitive Dysfunction; REM Sleep Behavior Disorder | interventions — 3-Iodobenzylguanidine; Iodine-123

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Myocardial 123I-MIBG scintigraphy imaging (Experimental): Subjects with with normal neurologic functioning, REM sleep without atonia, RBD, parkinsonism, cognitive impairment, or some combination of these will undergo myocardial 123I-MIBG scintigraphy imaging
  Interventions: Drug: meta-iodobenzylguanidine (MIBG) (123I); Diagnostic Test: 123I-MIBG scintigraphy

INTERVENTIONS:
Drug: meta-iodobenzylguanidine (MIBG) (123I) — 1 administration of 123I-MIBG for a single SPECT scan
  Other Names: 123I-MIBG
Diagnostic Test: 123I-MIBG scintigraphy — SPECT scan involving 123I-MIBG as the ligand

SUMMARY:
The purpose of the study is to investigate the use of a special radioactive drug called 123I-MIBG and myocardial MIBG scintigraphy. This scan may be able to help determine who may have a certain kind of neurologic disorder called Lewy Body Disease.

The overall purpose of this study is to correlate myocardial MIBG scintigraphy findings with clinical diagnosis. Myocardial MIBG scintigraphy imaging will be combined with other clinical, neuropsychological and neuroimaging findings to improve the prediction for underlying Lewy Body Disease.

DETAILED DESCRIPTION:
Lewy body disease (LBD) is one of the most common neurodegenerative diseases and second only to Alzheimer's disease in terms of prevalence, disability, and societal/financial burden. The clinical variability of LBD is striking, as it can manifest as Parkinson's disease (PD), PD with dementia (PDD), dementia with Lewy bodies (DLB), mild cognitive impairment (MCI), REM sleep behavior disorder (RBD), among other disorders. Considerable evidence now suggests that accumulation of the pathological protein and neuronal loss evolve over decades with RBD and/or MCI beginning years before developing overt DLB or PD.

This project investigates the utility of myocardial 123I-MIBG scintigraphy using a radioactive agent AdreView™ in participants with normal neurologic functioning, REM sleep without atonia, RBD, parkinsonism, cognitive impairment, or some combination of these. This scan may be able to help determine who may have underlying LBD.

Myocardial 123I-MIBG scintigraphy is considered as one of the most important imaging tests in the international diagnostic criteria of DLB, and it is widely used in European countries and Japan. Despite its globally recognized scientific importance, the use of AdreView™ and myocardial 123I-MIBG scintigraphy in DLB and associated disorders is not approved in the US. Currently, the FDA-approved indication of AdreView™ is limited to assessing specific cardiac function and detecting pheochromocytoma or neuroblastoma.

The overall purpose of this study is to correlate myocardial MIBG scintigraphy findings with clinical diagnosis. Myocardial MIBG scintigraphy imaging will be combined with other clinical, neuropsychological and neuroimaging findings to improve the detection of LBD. This study will help investigators learn the utility of myocardial 123I-MIBG scintigraphy in identifying LBD in the early course of the disease, and to prepare for clinical trials targeting LBD pathophysiology.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of one of the syndromes/diagnoses of interest using established criteria
* STMS score above 10
* No active medical disorder that could preclude participation
* Stable medication regimen over previous four weeks
* Absence of certain medications that could significantly impact the myocardial 123I-MIBG scintigraphy findings
* For those with dementia, caregiver that is with the patient at least 4 hours/day for at least 5 days per week
* For those with dementia, or severe parkinsonism, patient and caregiver willing and able to participate in all study-related procedures
* Patient is capable of giving informed consent, or if appropriate, has caregiver capable of giving consent on the subject's behalf.

Exclusion Criteria

* Does not fulfill criteria for any of the desired diagnoses
* Women with intact uterus and not post-menopausal unless pregnancy test performed at screening is negative
* Women who are pregnant or are breast-feeding an infant
* STMS score <10
* Active medical disorder that could preclude participation in this protocol

  * Hypersensitivity to the radioligand or iodine
  * Myocardial infarction or cerebral infarct over preceding year, stable or unstable angina, known symptomatic coronary artery disease
  * Renal disease viewed by the physician to be too severe to warrant myocardial 123I-MIBG scintigraphy imaging
  * History of significant alcohol or drug abuse
  * Any other medical disorder considered by the study physicians as inappropriate for enrollment in this protocol
* Patient or caregiver unwilling or unable to participate in all study-related procedures
* Caregiver is not with a patient with dementia or severe parkinsonism at least 4 hours/day for at least 5 days/week
* Patient or caregiver unwilling or unable to provide informed consent

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Correlate myocardial 123I-MIBG scintigraphy findings | 10 years
  Number of myocardial 123I-MIBG scintigraphy findings to correlate with clinical pathologic diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Boeve, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No